CLINICAL TRIAL: NCT05603832
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel Group Study of the Efficacy and Safety of a Single Administration of F14 for Postoperative Analgesia in Patients Undergoing Unilateral Total Knee Replacement
Brief Title: A Phase 3 Study of F14 for Management of Pain Following Total Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Arthritis Innovation Corporation (Industry)
Collaborators: Allucent (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 100-CIP02-P
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — N-nitrosobis(2,2,3,3,4,4,4-heptafluorobutyl)amine; Bupivacaine; Acetaminophen; Methocarbamol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- F14 + Multimodal Analgesia (Experimental)
  Interventions: Drug: F14; Drug: 0.25 % Bupivacaine HCl; Drug: Acetaminophen; Drug: Methocarbamol
- Multimodal Analgesia (Active Comparator)
  Interventions: Drug: 0.25 % Bupivacaine HCl; Drug: Acetaminophen; Drug: Methocarbamol

INTERVENTIONS:
Drug: F14 — 625 mg intra-articular sustained-release celecoxib
  Arms: F14 + Multimodal Analgesia
Drug: 0.25 % Bupivacaine HCl — Local anesthetic
Drug: Acetaminophen — Analgesic
Drug: Methocarbamol — Muscle relaxant

SUMMARY:
This is a Phase 3, randomized, double blind, multicenter study to evaluate the analgesic efficacy and safety of a single intra-articular dose of F14 (625 mg sustained release celecoxib) administered concurrent with multimodal analgesia in patients undergoing total knee replacement surgery, compared to multimodal analgesia alone.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or females indicated for primary, unilateral total knee replacement (TKR)
* Between 45-80 years of age inclusive at the time of signing the informed consent
* Capable of giving signed informed consent and complying with requirements and restrictions listed in the informed consent form (ICF) and in this protocol
* Body Mass Index (BMI) ≤ 40 kg/m2
* Medically stable as determined by the Investigator, based on physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG) findings, as well as medical history from patient and pre-study source documents from other care providers
* Absence of moderate to severe fixed flexion deformity
* Absence of moderate to severe varus or valgus deformity
* Minimum pre-operative flexion arc of 100 degrees
* Absence of steroid, hyaluronic acid, platelet rich plasma, or any other type of therapeutic injection(s) in the index knee within 3 months before scheduled surgery
* American Society of Anesthesiologists Physical Status Classification System (ASA-PSC) score ≤ 3
* Females of childbearing potential with a negative serum pregnancy test at screening, or males that have a partner who is a woman of child-bearing potential (WOCBP), who agree to employ adequate birth control measures for the full duration of the study.

Exclusion Criteria:

* Known allergy or hypersensitivity to active ingredient celecoxib, OR known allergy or hypersensitivity to sulfonamide antibiotics or sulfa containing drugs when an allergy to celecoxib is unknown
* Unwilling or unable to discontinue use of nonsteroidal anti-inflammatory drugs (NSAIDs) at least 7 days before study surgery and for 6 weeks following study surgery
* Unwilling or unable to discontinue use of medical or recreational marijuana or cannabidiol (CBD) at least 10 days before study surgery and for 3 months following study surgery
* Unwilling or unable to discontinue use of pregabalin, gabapentin or other drugs for neuropathic pain at least 7 days prior to study surgery and for 3 months following study surgery
* Unwilling or unable to discontinue opioid analgesics at least 7 days prior to surgery
* Has an allergy or contraindication to opioids or NSAIDs or acetaminophen
* Active or past infection in the index knee
* Total or partial knee arthroplasty in the contralateral knee < 6 months prior to study surgery
* Knee surgery (including cruciate ligament, cartilage or osteotomy) other than simple arthroscopy in either knee in the last 12 months (excluding contralateral total or partial knee replacement)
* Documented osteonecrosis within previous 12 months
* Prior or current presence of hardware in index knee other than screws from previous ligament repair that do not require manipulation or removal for TKR surgery
* Other planned major surgery within 12 months of study surgery
* Concurrent painful physical condition that is unrelated to the study knee (e.g., back, shoulder or contralateral knee pain) that will require analgesic treatment, such as NSAIDs or opioids, during study follow-up
* Current NRS pain intensity in the contralateral knee with a severity ≥ 4
* Current or historical evidence of any clinically significant disease or condition, especially cardiovascular, pulmonary or neurological, that, in the opinion of the Investigator, may increase the risk of surgery or complicate or affect the subject's study follow-up
* Suspected opioid abuse in the last 12 months with a score exceeding 5 on the DAST-10 questionnaire, and/or taking opioids ≥ 46 of the previous 90 days, and currently taking >90 mg in morphine milligram equivalents (MME) at least 5 days per week in the month prior to screening.
* History of alcohol abuse within previous 12 months (score of 4 on CAGE questionnaire)
* Anxiety Sensitivity Index (ASI) score >40
* Fear of Pain Score (FPQ-III) score >120
* Uncontrolled depression, mood or anxiety disorder (score exceeding 14 on PHQ-9 questionnaire)
* Participation or scheduled participation in another clinical study involving an investigational drug or device within one calendar month before screening or during study follow-up
* Current medical diagnosis or patient-reported seizure disorder
* Current peripheral neuropathy
* History of complex regional pain syndrome (CRPS)
* Diagnosis of clinically significant liver and/or renal abnormalities within previous 2 years
* Diagnosis of diabetes with HbA1c ≥7
* Current inflammatory arthritides (e.g., rheumatoid arthritis, lupus erythematosus, ankylosing spondylitis, psoriatic arthritis), or traumatic bone injuries within 12 months before scheduled surgery, except for clinically stable/non-active gout that does not affect the knee and does not interfere with walking
* Treatment with immunosuppressants within one calendar month of intervention. Also, antipsychotics, anticholinergics, or anticonvulsants within one calendar month of intervention unless stable dosage established for > one calendar month and does not plan to change during 3 month follow up
* Diagnosis of skin disorders including psoriasis, vascular insufficiency ulcers, and chronic venous stasis
* Subjects with sleep apnea associated with a history of postoperative delirium. If symptomatic sleep apnea is currently treated with continuous positive airway pressure (CPAP) or bilevel positive airway pressure (BIPAP), use must be continued post-operatively
* History of coronary or vascular stent placed within 3 months
* Had a malignancy in the last 12 months, except for non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix
* Positive urine drug screen for disallowed medication pre-operatively on day of study surgery
* Participation in active or pending personal injury or workers' compensation litigation related to index knee
* Any reason based on investigator clinical judgment, that subject may be non-compliant with respect to study obligations or assessments

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2024-08-23 (Actual)

PRIMARY OUTCOMES:
Time-weighted Area Under the Curve (AUC) of numeric rating scale (NRS) pain scores | 2 weeks

SECONDARY OUTCOMES:
Index knee range of motion (ROM) at 6 weeks | 6 weeks
Time-weighted AUC of NRS pain scores | 7 Days
Time-weighted AUC of NRS pain scores | 6 weeks
Proportion of subjects using opioid rescue medication at 2 weeks | 2 weeks
Time-weighted AUC of NRS pain scores | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Shive, PhD, Study Director — Arthritis Innovation Corporation
Locations (7):
- United States (7):
  - Woodland International Research Group, Little Rock, Arkansas
  - Phoenix Clinical Research, Tamarac, Florida
  - The Orthopedic Center, Tulsa, Oklahoma
  - HD Research - First Surgical Hospital, Bellaire, Texas
  - HD Research - Legent Orthopedic Hospital, Carrollton, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - CenExel JBR, Salt Lake City, Utah